CLINICAL TRIAL: NCT04464135
Title: Effect of Water Exchange Plus Acetic Acid Staining on the Detection of Flat Polyps During Screening and Surveillance Colonoscopy: a Multi-centered, Randomized Controlled Study.
Brief Title: Effect of Water Exchange Plus Acetic Acid Staining on the Detection of Flat Polyps During Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KY20200706-3
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Adenoma Colon
Keywords: Water exchange colonoscopy; Flat Polyps; Acetic Acid Staining

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WE+AA group (Experimental): Water containing 1% of AA was used during insertion of colonoscopy using water exchange method.
  Interventions: Other: acetic acid staining
- WE group (Active Comparator): Water exchange colonoscopy was used for standard screening or surveillance colonoscopy.
  Interventions: Other: Water exchange colonoscopy

INTERVENTIONS:
Other: acetic acid staining — The water exchange colonoscopy is used during insertion procedure, in which the water contains 1% acetic acid, and the liquid is absorbed during the withdrawal process for observation.
  Arms: WE+AA group
Other: Water exchange colonoscopy — The water exchange colonoscopy is used during insertion procedure, and the liquid is absorbed during the withdrawal process for observation.
  Arms: WE group

SUMMARY:
Our previous study (Am. J. Gastroenterol. 2017 04;112(4)) showed that water exchange (WE) colonoscopy was able to increase the detection of flat adenomas as well as overall ADR. We hypothesized that WE based whole-colon acetic acid（AA） staining might be useful to improve the detection of flat lesions compared with WE alone.

DETAILED DESCRIPTION:
Water exchange colonoscopy was performed as described previously (Am. J. Gastroenterol. 2017 04;112(4)). Patients were randomly allocated to WE group or WE+AA group. In WE+AA group, water containing 1% of AA was used during insertion of colonoscopy instead of water alone. A bottle of 20ml pure AA was placed abutting the water pump, which make it possible to keep patients blinded to group allocation. Endoscopist using a high-definition wide-angle Olympus or Fujinum colonoscope performed all of the colonoscopies, with a withdrawal time of at least 6 min. The observation was initially performed without the assistance of cap or the use of magnification or electronic staining (NBI, BLI, LCI or AFI et al.). Scopolamine butylbromide or glucogon was not routinely administrated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70
* Undergoing colonoscopy after standard bowel preparation

Exclusion Criteria:

* Known familial polyposis
* Small amount of feces or semi-solid stool in last rectal effluent
* Inflammatory Bowel Disease
* Lactated or pregnant women
* Unable to provide informed content

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of flat polyps per patient | 9 months
  average numbers of flat polyps, defined by Paris classification IIa/IIb/IIc, for each patient

SECONDARY OUTCOMES:
Overall ADR | 9 months
  Adenoma detection rate, defined as the proportion of subjects with at least one adenoma of any size, in each group.
Advanced ADR | 9 months
  Advanced adenoma detection rate. Advanced adenoma: any with 3 or more adenomas of any size, 1 or more large adenomas 1 cm, or 1 or more adenomas with villous architecture or highgrade dysplasia.
SSA/P detection rate | 9 months
  SSA/P detection rate, defined as the proportion of subjects with at least one sessile serrated adenoma/polyp (SSA/P) of any size, in each group.
Flat neoplasms located in proximal colon | 9 months
  Low-grade adenoma, adenoma with villous components, high-grade adenoma, noninvasive carcinoma, and invasive carcinoma in proximal colon
Adverse events | 9 months
  the rate of bleeding and perforation during colonoscopy procedure and abdominal pain, diarrhea, hematochezia and change of defecation habit Within one week.

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Xijing Hospital of Digestive Diseases
Locations (4):
- China (4):
  - Department of Gastroenterology, Second Affiliated Hospital, Lanzhou University, Lanzhou, Gansu
  - Department of Holistic Integrative Medicine, Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Department of Gastroenterology, Huaihe Hospital of Henan University, Kaifeng, Henan
  - Department of Gastroenterology, Shaanxi Second People's Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shibagaki K, Amano Y, Ishimura N, Yuki T, Taniguchi H, Fujita H, Kobayashi K, Kinoshita Y. Magnification endoscopy with acetic acid enhancement and a narrow-band imaging system for pit pattern diagnosis of colorectal neoplasms. J Clin Gastroenterol. 2015 Apr;49(4):306-12. doi: 10.1097/MCG.0000000000000148. PMID 24804989
- [Result] Jia H, Pan Y, Guo X, Zhao L, Wang X, Zhang L, Dong T, Luo H, Ge Z, Liu J, Hao J, Yao P, Zhang Y, Ren H, Zhou W, Guo Y, Zhang W, Chen X, Sun D, Yang X, Kang X, Liu N, Liu Z, Leung F, Wu K, Fan D. Water Exchange Method Significantly Improves Adenoma Detection Rate: A Multicenter, Randomized Controlled Trial. Am J Gastroenterol. 2017 Apr;112(4):568-576. doi: 10.1038/ajg.2016.501. Epub 2016 Dec 6. PMID 27922025
- [Result] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Result] Desai M, Sanchez-Yague A, Choudhary A, Pervez A, Gupta N, Vennalaganti P, Vennelaganti S, Fugazza A, Repici A, Hassan C, Sharma P. Impact of cap-assisted colonoscopy on detection of proximal colon adenomas: systematic review and meta-analysis. Gastrointest Endosc. 2017 Aug;86(2):274-281.e3. doi: 10.1016/j.gie.2017.03.1524. Epub 2017 Mar 29. PMID 28365356